CLINICAL TRIAL: NCT05765110
Title: SPEECH as Biomarker for Emotion, Movement and cOgnition in Parkinson's Disease
Acronym: EMO-SPEECH-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-01304
Record Dates: First submitted 2023-01-11; First posted 2023-03-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Speech; Emotion; Movement; Cognition; Biomarker; Automated speech analysis
MeSH Terms: conditions — Parkinson Disease; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson's disease patients with DBS (Experimental): All Parkinson's disease patients with bilateral deep brain stimulation (DBS) in the subthalamic nucleus
  Interventions: Other: Dopaminergic OFF drug state; Other: DBS OFF state; Other: Dopaminergic ON drug state; Other: DBS ON state
- Parkinson's disease patients without DBS (Experimental): All Parkinson's disease patients without bilateral deep brain stimulation (DBS) in the subthalamic nucleus
  Interventions: Other: Dopaminergic OFF drug state; Other: Dopaminergic ON drug state
- Healthy Controls (No Intervention): All healthy volunteers

INTERVENTIONS:
Other: Dopaminergic OFF drug state — Experiment will be performed without dopaminergic medication
  Arms: Parkinson's disease patients with DBS; Parkinson's disease patients without DBS
Other: DBS OFF state — Turning off the stimulation during experiment
  Arms: Parkinson's disease patients with DBS
Other: Dopaminergic ON drug state — Experiment will be performed with dopaminergic medication
  Arms: Parkinson's disease patients with DBS; Parkinson's disease patients without DBS
Other: DBS ON state — Experiment will be performed with stimulation (ON condition)
  Arms: Parkinson's disease patients with DBS

SUMMARY:
With this study, the investigators want to investigate whether computerized speech analysis can be used to reliably and objectively detect motor, emotional, and cognitive fluctuations in Parkinson's disease patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) affects mobility (motor function), thought processes (cognition) and mood (emotion). The language is one of the most complex programs in humans. It contains information about mobility, thinking and mood at the same time. These three levels of agility, thinking and mood are subject to spontaneous fluctuations and can be influenced by external stimuli such as pictures that induce emotions. In addition, these three levels are influenced on the one hand by Parkinson's disease itself, and on the other hand by its treatment with medication or with deep brain stimulation (DBS). For this reason, the investigators would like to investigate language in Parkinson's disease patients in a very detailed computerized way for motor, cognitive and emotional elements for better management of therapies.

With this study, the investigators want to investigate whether computerized speech analysis can be used to reliably and objectively detect fluctuations in motor, mood, and thinking in Parkinson's disease patients.

Even in healthy subjects, speech changes in a situational manner, due to which the investigators will also include healthy subjects as a control group.

ELIGIBILITY:
Patients with Parkinson's Disease

Inclusion Criteria:

* Written informed consent
* Idiopathic PD according to the Movement Disorders Society Criteria;
* Age of participants > 30 and ≤ 75 years;
* Treatment with or without bilateral deep brain stimulation in the subthalamic nucleus;
* Fluent in German or French

Exclusion Criteria:

* Dysarthria caused in addition by a condition other than PD (e.g. stroke, myasthenia);
* Clinical diagnosis of aphasia;
* Brain disease other than Parkinson's disease (e.g. atypical Parkinsonism, Alzheimer's disease, vascular dementia, multiple sclerosis, stroke, traumatic brain injury, epilepsy, etc.).
* Cognitive impairment (Montreal Cognitive Assessment (MoCa) < 24/30 points);
* Depression with acute suicidal ideation

Healthy Controls

Inclusion Criteria:

* Written informed consent
* Adults from 50-70 years old;
* Fluent in German or French

Exclusion Criteria:

* Diagnosis of Parkinson's disease;
* Cognitive impairment (Montreal Cognitive Assessment (MoCa) < 24/30 points);
* Suffering from brain disease (e.g. atypical Parkinsonism, Alzheimer's disease, vascular dementia, multiple sclerosis, stroke, traumatic brain injury, epilepsy, etc.);
* Clinical diagnosis of aphasia, dysarthria, and stuttering;
* Suffering from or diagnosed with psychiatric illnesses according to DSM-V criteria

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Part I: Changes from baseline in best acoustic speech variables to detect changes of dopaminergic and stimulation motor effect in Parkinson's disease patients | Visit 2 (< 3 months)
  A speech analyser software will allow extraction of basic motor acoustic speech features. The extracted variables that better index the dopaminergic medication or stimulation motor effect assessed with Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III - motor score [0-132 pts.] will be used as primary outcomes in this part. Higher scores in MDS-UPDRS part III means more severe motor symptoms.
Part II: Changes from baseline in best acoustic and linguistic speech variables to detect changes of dopaminergic and stimulation neuropsychological effect in Parkinson's disease patients | Visit 2 (< 3 months)
  A speech analyser software will allow extraction of basic acoustic speech features. For the linguistic domain several natural language variables will be extracted covering domains such as linguistic sense, coherence, and emotionality. The extracted variables that better index the dopaminergic medication or stimulation emotional effect assessed with Neuropsychiatric fluctuations scale (NFS) [0-60 pts.] will be used as primary outcomes in this part. Higher scores in NFS means more severe neuropsychiatric fluctuations.
Part III: Changes from baseline in best acoustic and linguistic speech variables to detect changes of dopaminergic and stimulation cognitive effect in Parkinson's disease patients | Visit 2 (< 3 months)
  A speech analyser software will allow extraction of basic acoustic speech features. For the linguistic domain several natural language variables will be extracted covering domains such as linguistic sense, coherence, and emotionality. The extracted variables that better index the dopaminergic medication or stimulation cognitive effect assessed with verbal fluency task will be used as primary outcomes in this part. Higher scores in Fluency task means better outcome.
Part III: Changes from baseline in best acoustic and linguistic speech variables to detect changes of dopaminergic and stimulation cognitive effect in Parkinson's disease patients | Visit 2 (< 3 months)
  A speech analyser software will allow extraction of basic acoustic speech features. For the linguistic domain several natural language variables will be extracted covering domains such as linguistic sense, coherence, and emotionality. The extracted variables that better index the dopaminergic medication or stimulation cognitive effect assessed with Stroop test will be used as primary outcomes in this part. Higher scores in Stroop test means worse outcome.

SECONDARY OUTCOMES:
Dyskinesia severity | At visit 1 (baseline) and visit 2 (< 3 months)
  Score on Marconi dyskinesia rating scale [0-28 pts.]. Higher scores in Marconi dyskinesia rating scale means more severe dyskinesia.
Momentary mood state | At visit 1 (baseline) and visit 2 (< 3 months)
  Score on Visual Analogue Mood Scale (VAMS) [0-100 pts.]. Higher scores in VAMS means better mood.
Momentary anxiety state | At visit 1 (baseline) and visit 2 (< 3 months)
  Score on Visual Analogue Anxiety Scale (VAAS) [0-100 pts.]. Higher scores in VAAS means more anxiety.
Bradyphrenia assessment | At visit 1 (baseline) and visit 2 (< 3 months)
  Score on Bradyphrenia scale [0-72 pts.]. Higher scores in Bradyphrenia scale means more severe bradyphrenia.

OTHER OUTCOMES:
Severity of non-motor aspects of experiences of Daily Living | < 2 weeks from the baseline visit
  Score on MDS-UPDRS parts I [0-52 pts.]. Higher scores in MDS-UPDRS-part I scale means more severe non-motor symptoms on experiences of Daily Living
Severity of motor aspects of experiences of Daily Living | < 2 weeks from the baseline visit
  Score on MDS-UPDRS parts II [0-52 pts.].Higher scores in MDS-UPDRS-part II scale means more severe motor symptoms on experiences of Daily Living
Severity of motor fluctuations | < 2 weeks from the baseline visit
  Score on MDS-UPDRS parts IV [0-24 pts.]. Higher scores in MDS-UPDRS-part IV scale means more severe motor fluctuations
Quality of life assessment | < 2 weeks from the baseline visit
  Score on Parkinson's Disease Questionnaire, 8 items (PDQ-8) [0-32 pts.]. Higher scores in PDQ-8 scale means worse quality of life
Dysarthria severity assessment | < 2 weeks from the baseline visit
  Score on Voice Handicap Index (VHI) [0-120 pts.]. Higher scores in VHI scale means more severe dysarthria (speech impairment)
Anxiety and depressive symptomatology | < 2 weeks from the baseline visit
  Score on Hospital Anxiety and Depression Scale (HADS) [0-60 pts.]. Higher scores in HADS scale means more severe anxiety and depressive symptoms
Apathetic symptomatology | < 2 weeks from the baseline visit
  Score on Starkstein Apathy Scale (SAS) [0-42 pts.]. Higher scores in SAS scale means more severe apathetic symptoms
Impulse-control disorders assessment | < 2 weeks from the baseline visit
  Score on Questionnaire for impulsive-compulsive disorders in Parkinson's Disease-Rating Scale (QUIP-RS) [0-112 pts.]. Higher scores in QUIP-RS scale means more severe impulsive-compulsive disorders

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krack, Prof., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Czech Technical University Prague, Prague, Czechia
- University Hospital Inselspital, Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No